CLINICAL TRIAL: NCT04955821
Title: Early Identification of Pathogens in Children With Respiratory Tract Infection by Mechanical Ventilation Using Metagenomics Next Generation Sequencing
Brief Title: Early Identification of Pathogens in Children With Respiratory Tract Infection by Mechanical Ventilation Using mNGS
Status: Not yet recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-22
Record Dates: First submitted 2021-07-05; First posted 2021-07-09 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: VAP - Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VAP group: Children with respiratory tract infection by mechanical ventilation
  Interventions: Diagnostic Test: mNGS diagnose of VAP

INTERVENTIONS:
Diagnostic Test: mNGS diagnose of VAP — This study is an observational study to evaluate the accuracy of pathogens in children with VAP tested by mNGS with no intervention. All patients from the cohort accept mNGS test and bacterial culture or virus PCR detection. A double sputum specimens are used for test.The reference standard is bacterial culture or virus PCR detection.

SUMMARY:
VAP（Ventilator-associated pneumonia）is the most common complication of mechanical ventilation in severely ill patients. VAP is defined as pneumonia occurring 48 hours after patients receive mechanical ventilation, including pneumonia occurring within 48 hours after extubation. It is one of the important causes of hospital-acquired infection, and the incidence of VAP in children on mechanical ventilation is about 10%, or 7/1000 days of mechanical ventilation, and the overall mortality is 10-24%.Research has so far explained the relationship between bacteria isolated from human biological samples and VAP pathogens. Most studies are limited to the level of bacterial species, and there are few reports on bacterial genotyping, and there is a lack of scientific basis for the pathogenesis of VAP caused by bacteria in ventilator pipeline. The aim of the study is to investigate pathogen of the sputum in deep respiratory tract of patients with mechanical ventilation in PICU by the means of second generation sequencing (NGS).

DETAILED DESCRIPTION:
Children receiving invasive mechanical ventilation in the intensive care unit (PICU) of the Pediatric Hospital of Fudan University will be included. Deep sputum samples were collected within 24 h and on day 5 of mechanical ventilation, respectively, and sent for NGS at the same time. Sputum etiology examination is performed with sputum culture blood free DNA test.

The basic clinical data of the children (age, sex, weight, PICU diagnosis and other basic information, as well as the time of start and end of invasive mechanical ventilation for basic diseases, Glasgow coma score (GCS score), 3rd generation pediatric mortality risk score III(Prism III score), CRP, PCT, white blood cell count and body temperature will be recorded。 Clinical data related to the use of glucocorticoids, antibiotics and other drugs as well as life support such as renal replacement therapy, extracorporeal membrane, lung oxygenation and other life support were collected. Time and method of diagnosis of VAP pathogens were collected.

By comparing sensitivity and specificity of NGS and conventional sputum specimens for detection of VAP, the clinical value of mNGS in VAP will be studied.

ELIGIBILITY:
Inclusion Criteria:

* The time of invasive mechanical ventilation was less than 24 h when admitted to PICU Total duration of invasive mechanical ventilation is over 5 days

Exclusion Criteria:

* Participants in other clinical trials in the same period No Informed Consent signed

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children receiving invasive mechanical ventilation in PICU
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The accuracy of mNGS diagnosis in identification of pathogens in children with VAP. | within 28 days after being discharged from PICU
  The accuracy of combined diagnosis includes sensitivity and specificity. The reference standard test ( bacterial culture or virus PCR detection) and mNGS diagnosis are conducted in the cohort of pediatric children diagnosed of VAP

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Lu, doctor, Principal Investigator — Children's Hospital of Fundan University

IPD SHARING:
Plan to Share IPD: No